CLINICAL TRIAL: NCT04449978
Title: TARGet Kids! COVID-19 Study of Children and Families
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Catherine Birken, Senior Scientist, The Hospital for Sick Children
Other Study IDs: 1000069701
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Coronavirus; COVID-19; Virus; Family and Household; Infection Viral
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal swab samples, dried blood spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The novel coronavirus (COVID-19) was declared a global pandemic in March 2020. Early research suggests that children are no more susceptible to COVID-19 infection than adults and that children with confirmed COVID-19 have generally presented with milder symptoms. However, the impact of COVID-19 among Canadian children remains unclear. The prevalence of COVID-19 in children in Canada is currently unknown and no published research exists regarding the risk factors of COVID-19 in children or its potential long-term health effects on physical health or development. Using TARGet Kids!, Canada's largest children's cohort study with over 11,000 children involved, the researchers will conduct a longitudinal observational study aimed to evaluate the cumulative incidence of COVID-19 in children and parents; differences among infected and uninfected children in terms of age, sex, and income; risk factors of COVID-19; and longer term health effects of COVID-19 among children. Given the rapid spread of COVID-19 and the unknown health effects of the virus in children, research must be conducted to determine the extent of infections of COVID-19 in children, disease severity, risk factors for infection, and how the virus affects children as they become older.

DETAILED DESCRIPTION:
The novel coronavirus (COVID-19) was declared a global pandemic in March 2020. Early research has suggested that children may experience less severe clinical symptoms than adults, and infected children with minimal or no symptoms may be an underrecognized source of community disease transmission. COVID-19 infections in children were occurring very early in the epidemic but the impact of COVID-19 infection among children remains unclear. The number of COVID-19 infections in children and parents in Canada is unknown and studies have not evaluated the symptom severity of COVID-19 in children and parents, risk factors for infection and severe disease, and whether current preventive efforts are effective. Using TARGet Kids!, Canada's largest children's cohort study, the researchers will conduct an observational study to evaluate key epidemiological characteristics of COVID-19 among parents and children, as well as to determine the spectrum of disease severity, seroprevalence, risk factors for COVID-19 infection and severe disease, effectiveness of social isolation recommendations, risk to family members with a COVID-19 infected family member, and potential new strategies to prevent COVID-19 infection and minimize disease severity. Parents of 1082 existing TARGet Kids! participants will be asked to provide a nasal swab from themselves and their child during the pandemic in addition to a respiratory tract symptom checklist. Preventive efforts (e.g. social distancing), parent-reported illness, laboratory-confirmed infections and healthcare encounters (e.g. emergency department visits, hospitalizations and ICU care) will be measured. Children will subsequently be followed through the TARGet Kids! cohort study over the next 6 months and long term, with interim analyses at 3 months. By understanding every stage of COVID-19 infection from prevention to transmission in the community and home, to outpatient and hospital care utilization, the researchers will rapidly develop new interventions to prevent COVID-19 transmission and minimize disease severity among children and their families. Descriptive statistics will be used to determine the prevalence of COVID-19 in healthy children.

ELIGIBILITY:
Inclusion Criteria:

* Families with existing participants of the TARGet Kids! cohort with children between the ages of 0-16 years.

Exclusion Criteria:

* Families who are not participating in the TARGet Kids! cohort or participating families with no children within the age of eligibility.

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will be a prospective longitudinal observational study embedded within the TARGet Kids! cohort study, an ongoing longitudinal observational study enrolling healthy age 0-5 years who receive primary healthcare and following them until adolescence and early adulthood.
Sampling Method: Non-Probability Sample
Enrollment: 1145 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative Incidence of COVID-19 | 12 months
  To evaluate the cumulative incidence of laboratory-confirmed COVID-19 among healthy children and parents in Toronto, Canada

SECONDARY OUTCOMES:
Risk Factors for COVID-19 | 12 months
  To determine the risk factors for COVID-19 infection in children and parents to inform preventive interventions
Parent-reported probable case definition of COVID-19 | 12 months
  To determine the cumulative incidence of parent-reported probable case definition of COVID-19 among children and parents.
Dynamics of COVID-19 | 12 months
  To determine the dynamics of COVID-19 infection using a susceptible-infected-recovered (SIR) multi-state model.
Risk to family members | 12 months
  To determine the risk to family members with a laboratory-confirmed COVID-19 infected family member.
Severity of COVID-19 | 12 months
  To determine the severity of laboratory-confirmed COVID-19 in healthy children and parents
Longer term effects of COVID-19 on physical health | 12 months
  To determine the longer term effects of COVID-19 infection in healthy children and parents on physical health
Longer term effects of COVID-19 on mental health | 12 months
  To determine the longer term effects of COVID-19 infection in healthy children and parents on mental health
Longer term effects of COVID-19 on child development | 12 months
  To determine the longer term effects of COVID-19 infection in healthy children and parents on child development
Longer term effects of COVID-19 on family functioning | 12 months
  To determine the longer term effects of COVID-19 infection in healthy children and parents on family functioning
Longer term effects of COVID-19 on health behaviours | 12 months
  To determine the longer term effects of COVID-19 infection in healthy children and parents on health behaviours
Longer term effects of COVID-19 on healthcare utilization | 12 months
  To determine the longer term effects of COVID-19 infection in healthy children and parents on healthcare utilization
Effects of preventive measures on infection | 12 months
  To determine the effect of preventive measures on COVID-19 infection
Effects of preventive measures on physical health | 12 months
  To determine the effect of preventive measures on physical health
Effects of preventive measures on mental health | 12 months
  To determine the effect of preventive measures on mental health
Effects of preventive measures on child development | 12 months
  To determine the effect of preventive measures on child development
Effects of preventive measures on family functioning | 12 months
  To determine the effect of preventive measures on family functioning
Effects of preventive measures on health behaviours | 12 months
  To determine the effect of preventive measures on health behaviours
Effects of preventive measures on healthcare utilization | 12 months
  To determine the effect of preventive measures on healthcare utilization

CONTACTS AND LOCATIONS:
Overall Officials: Catherine S Birken, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - St Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.